CLINICAL TRIAL: NCT02278796
Title: A Randomized Phase II Trial Comparing BeEAM With BEAM as Conditioning Regimen for Autologous Stem Cell Transplantation (ASCT) in Lymphoma Patients (BEB-trial)
Brief Title: A Trial Comparing the Two High-dose Chemotherapies BeEAM and BEAM Given Before Autologous Stem Cell Transplantation (ASCT) in Lymphoma Patients (BEB-trial)
Acronym: BEB
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Hanusk Krankenhaus Wien (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEB-Trial; 2014-003629-16 (EudraCT Number)
Record Dates: First submitted 2014-10-15; First posted 2014-10-30 (Estimated); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell
Keywords: Diffuse large B-cell lymphomas (DLBC); Follicular lymphomas (FL); Mantle cell lymphomas (MCL)
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- BeEAM (Experimental): Chemotherapy regimen consisting of bendamustine intravenously on days -7 and -6 at 200 mg/m2; cytarabine, 400 mg/m2 intravenously daily from day -5 to day-2; etoposide, 200 mg/m2 intravenously daily from day -5 to day -2; and melphalan, 140 mg/m2 intravenously on day -1 before reinfusion of autologous stem cells
  Interventions: Drug: BeEAM
- BEAM (Active Comparator): Chemotherapy regimen with carmustine (BCNU) 300 mg/m2 on day -6, cytarabine, 400 mg/m2 intravenously daily from day -5 to day-2; etoposide, 200 mg/m2 intravenously daily from day -5 to day -2; and melphalan, 140 mg/m2 intravenously on day -1 before reinfusion of autologous stem cells
  Interventions: Drug: BEAM

INTERVENTIONS:
Drug: BeEAM — Chemotherapy regimen consisting of bendamustine intravenously on days -7 and -6 at 200 mg/m2; cytarabine, 400 mg/m2 intravenously daily from day -5 to day-2; etoposide, 200 mg/m2 intravenously daily from day -5 to day -2; and melphalan, 140 mg/m2 intravenously on day -1 before reinfusion of autologous stem cells
  Arms: BeEAM
Drug: BEAM — Chemotherapy regimen with carmustine (BCNU) 300 mg/m2 on day -6, cytarabine, 400 mg/m2 intravenously daily from day -5 to day-2; etoposide, 200 mg/m2 intravenously daily from day -5 to day -2; and melphalan, 140 mg/m2 intravenously on day -1 before reinfusion of autologous stem cells
  Arms: BEAM

SUMMARY:
In the treatment of patient with lymphoma the most common high-dose chemotherapy regimen used prior to autologous transplantation (ASCT) is the BEAM regimen. It consists of four chemotherapy drugs together (BCNU, etoposide, cyclophosphamide, melphalan), whose initial letters are grouped together for BEAM regimen. One of the most common organ damage this intensive treatment is caused by the drug BCNU; it involves a lung injury, which manifests itself in the months after ASCT with increasing shortness of breath and cough, and can result in pulmonary fibrosis. The drug bendamustine is used successfully in different lymphoma types, and its efficacy in lymphoma therapy is well documented. Moreover bendamustine doesn't cause lung injury. Initially experience with bendamustine instead of BCNU - in the so-called BeEAM scheme - shows that this scheme is quite effective and well tolerated, without lung injury. In BeEAM scheme therefore bendamustine replace the BCNU, while the other three drugs are administered in the same dosage and order. The aim of the present study conducted at four centers (Bern and Zurich in Switzerland, Vienna and Linz in Austria) is to compare these two high-dose chemotherapy schemas and to show that the BeEAM scheme causes significantly less lung injury than the BEAM regimen.

DETAILED DESCRIPTION:
Background

High-dose chemotherapy (HDCT) followed by autologous stem cell transplantation (ASCT) is considered the treatment of choice for relapsed/refractory lymphomas. On the basis of the results of the PARMA study group trial, high-dose chemotherapy followed by ASCT has become the standard of care for patients with relapsed, chemo-sensitive aggressive lymphoma and it is the treatment of choice in patients relapsing with follicular lymphoma and Hodgkin's disease. The BEAM (BCNU, etoposide, cyclophosphamide, melphalan) chemotherapy regimen is the most frequently used conditioning regimen since more than thirty years. Toxic pneumonia with interstitial infiltration and impairment of the diffusion capacity of the lung is a recognized complication of HDCT regimens containing BCNU. Recently, it has been shown that the EAM regimen (thus omitting BCNU) is not sufficient to obtain equal response rates if compared with BEAM and poorer disease control resulted in impaired disease-free survival (DFS). Thus, it might be detrimental for patients just to eliminate BCNU without an appropriate substitution. Replacing BCNU by Bendamustine with its potential to eradicate residual or treatment-resistant lymphoma cells could be a promising clinical approach and should be investigated in a randomized phase II clinical trial comparing standard BEAM with BeEAM. Bendamustine combines the alkylating activity of the mustard group with the antimetabolite activity of the purine analogue and was studied in several entities of B-cell neoplasms and demonstrated significantly superior efficacy compared with standard therapies in the treatment of relapsed chronic lymphocytic leukemia (CLL) and indolent NHL and myeloma. The BRIGHT study confirmed the non-inferiority of a immunochemo-therapy with Rituximab-Bendamustine when compared with R-CHOP or Rituximab, Cyclophosphamide, Vincristine, Prednisone (R-CVP) in indolent lymphoma or mantle cell lymphoma. Recently, Visani et al have shown that Bendamustine, coupled with fixed doses of Etoposide, Cytarabine, and Melphalan (ie, BeEAM) in the conditioning regimen for ASCT for resistant/relapsed lymphoma (HD and NHL) patients is highly active and resulted in promising results concerning safety and efficacy. No treatment mortality was observed and no relevant pulmonary toxicity was seen. Non-hematological toxicity was moderate, and most prominent toxicities were gastroenteritis grade 3 to 4 in 34% and mucositis grade 3 to 4 in 35%, respectively. No grade 3 to 4 cardiac toxicity or toxic pneumonia was observed. Engraftment was rapid and trilinear, and stable hematopoiesis was observed. BeEAM was very effective, with 81% of patients in complete response after a median observation time of 18 months. A recent update of this study showed that at 41 months still 72% of the patients are still in complete remission and the 3-year performance status (PS) was 75%. Four patients showed a first remission ever with the Bendamustine containing regimen. In 35 patients treated at the Vienna centre according to the Visani BeEAM protocol, these encouraging data of Visani et al could be reproduced; similar toxicities and rapid and stable engraftment were observed. Finally, the combination of Bendamustine with sequential application of high-dose Cytarabine was reported to improve the response rates in relapsing lymphomas. In conclusion, it seems promising to integrate Bendamustine in myeloablative regimens in ASCT, but a randomized clinical trial is lacking so far.

Objective

Replacing the chemotherapeutic drug BCNU by Bendamustine within the four-drug chemotherapy regimen BEAM reduces the occurrence of early and late pulmonary toxicity in lymphoma patients undergoing high-dose chemotherapy with autologous stem cell transplantation. Primary Objective: To show a clinically meaningful reduction of lung toxicity - defined as a a decrease of the diffusion capacity of the lung for carbon monoxide (DLCO) by 20% or more from baseline before ASCT - from 25% of patients in the BEAM group to 4% of patients in the BeEAM group at 3 months after ASCT. Use Dinakara equation for adjusting DLCO for hemoglobin. Secondary Objectives: Acute and late toxicity/adverse events (CTCAE 4.0). Hematologic recovery and engraftment after 3 months. Early and late lung toxicity Cardiac assessment by ECHO/ECG and quality of life before,3 and 12 months after ASCT. Overall survival and progression free survival after 12 months and then yearly as routine follow-up assessments.

Methods

Two high-dose chemotherapy regimens (BeEAM versus BEAM) used for conditioning treatment before autologous stem cell transplantation will be compared in a 1:1 randomization. The experimental arm is the BeEAM regimen. The BEAM regimen is the control treatment. Lung toxicity will be assessed by spiroergometry at the 60% level of maximum exercise capacity, as well as by assessing the diffusion capacity of the lung for carbon monoxide (DLCO). This analysis will be performed before ASCT, as well as 3 months and 12 months after ASCT. Patients will be assessed for cardio-pulmonary toxicity before ASCT, as well as 3 and 12 months after ASCT. Thereafter, patient follow-up will be performed clinically once per year.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Chemosensitive diffuse large B-cell lymphomas (DLBCL), follicular lymphomas (FL), and mantle cell lymphomas (MCL) in first or second remission
* Aged between 18 years and 75 years
* Neutrophils ≥ 1000/μl; Platelets ≥ 100 x 109/L

Exclusion Criteria

* Acute uncontrolled infection
* Clinically significant concomitant disease states
* Hematopoietic cell transplantation comorbidity index (HCT-CI) > 5
* Previous or concurrent malignant disease with the exception of basalioma/spinalioma of the skin or early-stage cervix carcinoma
* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Major coagulopathy or bleeding disorder
* Major surgery less than 30 days before start of treatment
* Contraindications to the class of drugs under study, known hypersensitivity or allergy to class of drugs or the investigational product
* Women who are pregnant or breast feeding; Women with the intention to become pregnant during the course of the study
* Lack of safe contraception
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pabst, Prof Dr. med, Study Chair — Department for Medical Oncology University Hospital/Inselspital; Felix Keil, Prim. Univ. Prof. Dr, Principal Investigator — Hanusch Krankenhaus Wien
Locations (4):
- Austria (2):
  - Krankenhaus der Elisabethinen Linz, Linz
  - Hanusch Krankenhaus Wien, Vienna
- Switzerland (2):
  - Department for Medical Oncology University Hospital/Inselspital, Bern
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Visani G, Malerba L, Stefani PM, Capria S, Galieni P, Gaudio F, Specchia G, Meloni G, Gherlinzoni F, Giardini C, Falcioni S, Cuberli F, Gobbi M, Sarina B, Santoro A, Ferrara F, Rocchi M, Ocio EM, Caballero MD, Isidori A. BeEAM (bendamustine, etoposide, cytarabine, melphalan) before autologous stem cell transplantation is safe and effective for resistant/relapsed lymphoma patients. Blood. 2011 Sep 22;118(12):3419-25. doi: 10.1182/blood-2011-04-351924. Epub 2011 Aug 3. PMID 21816830
- [Result] Loke J, Ward J, Mahendra P, Chaganti S, Malladi R. Outcomes of EAM conditioned autologous haematopoietic SCT for lymphoma. A matched pairs retrospective single-centre study analysis. Bone Marrow Transplant. 2013 Nov;48(11):1486-7. doi: 10.1038/bmt.2013.90. Epub 2013 Jun 10. No abstract available. PMID 23749106
- [Result] Alessandrino EP, Bernasconi P, Colombo A, Caldera D, Martinelli G, Vitulo P, Malcovati L, Nascimbene C, Varettoni M, Volpini E, Klersy C, Bernasconi C. Pulmonary toxicity following carmustine-based preparative regimens and autologous peripheral blood progenitor cell transplantation in hematological malignancies. Bone Marrow Transplant. 2000 Feb;25(3):309-13. doi: 10.1038/sj.bmt.1702154. PMID 10673703
- [Result] Flinn IW, van der Jagt R, Kahl BS, Wood P, Hawkins TE, Macdonald D, Hertzberg M, Kwan YL, Simpson D, Craig M, Kolibaba K, Issa S, Clementi R, Hallman DM, Munteanu M, Chen L, Burke JM. Randomized trial of bendamustine-rituximab or R-CHOP/R-CVP in first-line treatment of indolent NHL or MCL: the BRIGHT study. Blood. 2014 May 8;123(19):2944-52. doi: 10.1182/blood-2013-11-531327. Epub 2014 Mar 3. PMID 24591201
- [Result] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Derived] Keil F, Muller AMS, Berghold A, Riedl R, Buxhofer-Ausch V, Schuster J, Vorburger C, Bohm A, Panny M, Nosslinger T, Greil R, Samaras P, Bencker C, Rutti M, Pabst T. BendaEAM versus BEAM as conditioning regimen for ASCT in patients with relapsed lymphoma (BEB): a multicentre, randomised, phase 2 trial. EClinicalMedicine. 2023 Nov 19;66:102318. doi: 10.1016/j.eclinm.2023.102318. eCollection 2023 Dec. PMID 38024477

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BeEAM | BEAM
Started | 53 | 55
Completed | 51 | 52
Not Completed | 2 | 3
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BeEAM | BEAM | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 55 | 108
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (1.1) | 51.9 (1.1) | 51.85 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 36 | 39 | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 19 | 20 | 39
  Switzerland | 34 | 35 | 69

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Clinically Meaningful Reduction in Lung Toxicity, Defined as a Reduction of the Diffusion Capacity of the Lung for Carbon Monoxide (DLCO) by at Least 20%.
Description: Number of patients with a clinically meaningful reduction in lung toxicity, defined as a reduction of the diffusion capacity of the lung for carbon monoxide (DLCO) by at least 20%. DLCO measured in mmol/min/kPA
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 51 | 52
Participants | 8 | 11

2. Secondary Outcome: Acute Toxicity/Adverse Events (CTCAE4)
Description: Overall number of adverse events grade 3-5 at ≤ 35 days after ASCT (CTCAE4)
Time Frame: ≤ 35 days
Measure: Number; unit: Events
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 53 | 55
Events | 19 | 17

3. Secondary Outcome: Hematologic Recovery and Engraftment (ANC)
Description: Hematologic recovery measured as median time (days) to ANC >0.5 × 10 ^9/l
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 52 | 54
days | 10 [10 to 11] | 10 [10 to 11]

4. Secondary Outcome: Percentage of Patients With Overall Survival
Description: Percentage of patients alive after autologous stem cell transplantation after one year
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 53 | 55
percentage of participants | 92.3 [80.8 to 97] | 88.6 [76.3 to 94.7]

5. Secondary Outcome: Late Toxicity/Adverse Events (CTCAE4)
Description: Number of events grade 3-5 AE at 1 year after ASCT (CTCAE4)
Time Frame: Continuously up to 1 year
Measure: Number; unit: events
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 47 | 42
events | 22 | 6

6. Secondary Outcome: Hematologic Recovery and Engraftment (PLT)
Description: Hematologic recovery neasured as median time (days) to PLT >20 × 10^9/l
Time Frame: 100 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BeEAM | BEAM
Number analyzed (Participants) | 51 | 53
days | 12 [11 to 14] | 12 [10 to 17]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | BeEAM | BEAM
All-Cause Mortality (participants affected / at risk) | 4/53 | 6/55
Serious Adverse Events (participants affected / at risk) | 6/53 | 6/55
Other Adverse Events (participants affected / at risk) | 31/53 | 25/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeEAM (N=53) | BEAM (N=55)
Infection (Infections and infestations) | 6 (6) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BeEAM (N=53) | BEAM (N=55)
Gastrointestinal disorders (Gastrointestinal disorders) | 31 (31) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT02278796/Prot_SAP_000.pdf